CLINICAL TRIAL: NCT06095180
Title: Comparison of Efficacy of Ultrasound-Guided Steroid Injection and Dry Needling in Piriformis Muscle Syndrome
Brief Title: Comparison of Ultrasound-guided Steroid Injection and Dry Needling in Piriformis Muscle Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Piriformis Muscle Syndrome
Keywords: piriformis syndrome; steroid injection; dry needling; exercise
MeSH Terms: conditions — Piriformis Muscle Syndrome; Motor Activity | interventions — Adrenal Cortex Hormones; Dry Needling; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be evaluated by an independent physiatrist, blinded for the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- corticosteroid group (Active Comparator): In the steroid group, 4 mL lidocaine 2% + 1 mL betamethasone injection will be administered under ultrasound guidance and conventional treatment will be given (conventional treatment includes piriformis stretching exercises. It will be stated that patients should do 2 sets a day and each set should be 10 repetition)
  Interventions: Other: corticosteroid injection
- dry needling group (Active Comparator): In the dry needling group, a total of 3 sessions of dry needling will be performed once a week using a 0.60×100 mm sterile needle under ultrasound guidance and conventional treatment will be given ((conventional treatment includes piriformis stretching exercises. It will be stated that patients should do 2 sets a day and each set should be 10 repetition)
  Interventions: Other: dry needling
- control group (Other): The conventional treatment group (control group) will be given piriformis stretching exercises including hip and knee flexion, hip abduction and external rotation in the supine position. It will be stated that patients should do 2 sets a day and each set should be 10 repetitions.
  Interventions: Other: exercise

INTERVENTIONS:
Other: corticosteroid injection — In the steroid group, 4 mL lidocaine 2% + 1 mL betamethasone injection will be administered under ultrasound guidance and conventional treatment will be given (conventional treatment includes piriformis stretching exercises. It will be stated that patients should do 2 sets a day and each set should be 10 repetition)
  Arms: corticosteroid group
Other: dry needling — In the dry needling group, a total of 3 sessions of dry needling will be performed once a week using a 0.60×100 mm sterile needle under ultrasound guidance and conventional treatment will be given ((conventional treatment includes piriformis stretching exercises. It will be stated that patients should do 2 sets a day and each set should be 10 repetition)
  Arms: dry needling group
Other: exercise — The conventional treatment group (control group) will be given piriformis stretching exercises including hip and knee flexion, hip abduction and external rotation in the supine position. It will be stated that patients should do 2 sets a day and each set should be 10 repetitions.
  Arms: control group

SUMMARY:
The aim of this study is to to compare its effectiveness ultrasound-guided steroid injection, dry needling treatments and exercises in patients diagnosed with piriformis syndrome.

DETAILED DESCRIPTION:
Piriformis syndrome is a painful entrapment neuropathy caused by compression of the sciatic nerve under the piriformis muscle. The most common cause is myofascial pain syndrome. There is no gold standard treatment for piriformis syndrome. The main purpose of treatment methods is to reduce local pain, muscle tension and spasm. This work; it will contribute to the literature by comparing steroid, dry needling and exercise treatments in patients with piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60,
2. Hip pain for ≥1 month
3. Local piriformis pain with prolonged sitting (>20 minutes) and increased sensitivity
4. Patients with suspected piriformis syndrome based on clinical maneuvers
5. Signing and informed consent from showing consent to participate in the study

Exclusion Criteria:

1. Hip surgery
2. Lumbar disc disease
3. History of inflammatory hip disease
4. Medical treatment for pain is started
5. Neurological deficit
6. Breastfeeding or pregnant
7. Allergy to local anesthetic
8. Use of anticoagulants
9. Body mass index >35
10. Active psychiatric illness
11. Uncontrolled hypertension and diabetes mellitus disease
12. Noncompensated chronic lung/heart/renal failure
13. History of vascular/tumoral disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-28 (Estimated); Primary Completion 2024-08-26 (Estimated); Study Completion 2024-08-26 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) (Sitting) | at baseline and change from baseline VAS (sitting) at 4 weeks and 12 weeks
  Average hip pain intensity in a sitting position over the past 24 hours, a visual analog scale. (VAS; ranging from 0 to 10, 0 = no pain and 10 = worst possible pain)
Visual Analog Scale (VAS) (Resting) | at baseline and change from baseline VAS (resting) at 4 weeks and 12 weeks
  Average hip pain intensity at rest over the past week is a visual analog scale. (VAS; ranging from 0 to 10, 0 = no pain and 10 = worst possible pain)
Visual Analog Scale (VAS) (Movement) | at baseline and change from baseline VAS (movement) at 4 weeks and 12 weeks
  Average hip pain intensity during movement over the past 1 week is a visual analog scale. (VAS; ranging from 0 to 10, 0 = no pain and 10 = worst possible pain)

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | at baseline and change from baseline ODI at 4 weeks and 12 weeks
  ODI includes questions regarding pain severity, sexual function, sleep quality and personal care, ability to work, sit, walk, lift, stand and travel. Total score ranges from 0-50, with higher scores indicating more injury.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Şimşek Yağlıoğlu, MD, Principal Investigator — Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital